CLINICAL TRIAL: NCT02495220
Title: Subtenon Versus Intravenous Dexmedetomidine for Postoperative Analgesia and Vomiting Control in Infantile Cataract Surgery
Brief Title: Efficacy of Dexmedetomidine for Postoperative Analgesia in Infantile Cataract Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, jehan ahmed sayed, assistant professor in anesthesia and intensive care department,faculty of medicine assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00008711068
Record Dates: First submitted 2015-07-03; First posted 2015-07-13 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Pain; Postoperative Vomiting
Keywords: dexmedetomidine; subtenon anesthesia; postoperative pain; pov
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- subtenon block Group (SB) (Experimental): received SB block with 0.05 mL/kg of 0.5%bupivacaine and 0.5µ/kg dexmedetomidine mixture
  Interventions: Drug: SB dexmedetomidine bupivacaine block
- intravenous dexmedetomidine Group(IV) (Experimental): received 1µ/kg IV dexmedetomidine after induction of anesthesia
  Interventions: Drug: intravenous dexmedetomidine

INTERVENTIONS:
Drug: SB dexmedetomidine bupivacaine block — SB block with 0.05 mL/kg of 0.5%bupivacaine and 0.5µ/kg dexmedetomidine mixture
  Arms: subtenon block Group (SB)
Drug: intravenous dexmedetomidine — received 1µ/kg IV dexmedetomidine
  Arms: intravenous dexmedetomidine Group(IV)

SUMMARY:
The purpose of the present study was to evaluate the efficacy and safety of subtenon block (SB)anesthesia with dexmedetomidine in combination with bupivacaine versus intravenous dexmedetomidine for postoperative analgesia and emesis control in infants undergoing cataract surgery.

DETAILED DESCRIPTION:
In this prospective, randomized, controlled, double blind trial eighty ASA physical status grade I and II infants (1-12month) undergoing elective cataract surgery in one eye under general anesthesia were studied. Infants were randomly allocated to one of the two groups: subtenon block Group (SB) with dexmedetomidine (n =40) or intravenous dexmedetomidine Group (IV) (n =40). After securing the airway, infants in Group (SB) received SB block with 0.05 mL/kg of 0.5%bupivacaine and 0.5µ/kg dexmedetomidine mixture, whereas infants in Group (IV) received 1µ/kg IV dexmedetomidine after induction of anesthesia. Surgery started after 5 min of study drug administration. Postoperative assessment for number of infants requiring rescue analgesia and rescue antiemetics was the primary outcome. CRIES pain scale score , vomiting scale score during4-h study period, incidence of oculocardiac reflex and any surgical difficulty were the Secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status grade I and II infants (1-12month).
2. undergoing elective cataract surgery in one eye under general anesthesia.

Exclusion Criteria:

1. infection of the orbit,
2. increased intraocular pressure(IOP),
3. history of allergy to local anesthetics,
4. history of previous eye surgery,
5. cardiovascular or clotting disorders,
6. full stomach,inner ear disorders or other conditions predisposing to vomiting
7. airway abnormalities
8. compromised sclera.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative assessment for number of infants requiring rescue analgesia and rescue antiemetics | 4 hours postoperatively
  by analysis for number of infants withCRIES pain scale score >3
postoperative CRIES pain scale score | 4 hours postoperatively
  (0-2 for each parameter)

SECONDARY OUTCOMES:
vomiting scale score | 4 hours postoperative
  a numeric rank score, where 0= no vomiting 1=vomited once and 2=vomited twice or more
Number of oculocardiac reflex(OCR)events(acute reduction in heart rate of >20%). | intraoperative period
  by analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Univeristy Hospital, Asyut, Egypt